CLINICAL TRIAL: NCT00004234
Title: A Comparison of Acute Oral Mucositis Between Morning and Afternoon Radiotherapy in Patients Receiving Radiation Treatment for Cancer of the Head and Neck
Brief Title: Oral Mucositis in Patients Receiving Radiation Therapy for Cancer of the Mouth, Pharynx, or Larynx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: HN3; CAN-NCIC-HN3 (Other: PDQ); CDR0000067478 (Other: PDQ)
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Cancer; Oral Complications
Keywords: oral complications; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I squamous cell carcinoma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: management of therapy complications
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation therapy at different times of the day may affect the chance of developing side effects such as mucositis.

PURPOSE: Randomized phase III trial to compare the incidence of mucositis in patients who have cancer of the mouth, pharynx, or larynx, who are receiving radiation therapy in either the morning or afternoon.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the toxicity of radiotherapy to the oral mucosa delivered in the morning or in the late afternoon in patients with squamous cell carcinoma of the oral cavity, pharynx (oro/hypo/naso), or larynx who will receive radiation treatment to a significant part of the oral and/or oropharyngeal mucosa.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, intended smoking behavior during therapy (smoking vs nonsmoking), and planned total radiotherapy dose.

Patients are randomized to receive radiotherapy once daily, 5 days a week, at one of two of the following times of the day:

* Arm I: Patients receive radiotherapy between 8 and 10 AM (local time).
* Arm II: Patients receive radiotherapy between 4 and 6 PM (local time). Treatment continues for 5-8 weeks, depending on planned total radiotherapy dose, in the absence of unacceptable toxicity or disease progression.

Toxicity is assessed at baseline, at the first fraction of radiotherapy, weekly during treatment, weekly until mucositis has peaked and is improving, and then every 2 weeks until mucositis has improved to less than grade 2.

Quality of life is assessed at baseline, weekly during treatment and until toxicity has peaked and is improving, every 2 weeks until toxicity is less than grade 2 mucositis, and then at each follow-up visit until week 24.

Patients are followed at weeks 2-3, 6-8, 12, and 24 and then annually for 3 years.

PROJECTED ACCRUAL: A total of 216 patients (108 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, pharynx (oropharynx, hypopharynx, or nasopharynx), or larynx eligible for radical radiotherapy

  * TX, T1-4, NX, N0-3, M0
  * Directly visible area of mucosa including 2 or more protocol specified anatomical locations in the radical target volume

    * At least 6 cm^2 in area irrespective of shape
  * No M1 disease
* Intention to deliver radiotherapy to a radical dose without chemotherapy
* May have had surgical resection of the primary or neck nodes

  * Postoperative macroscopic or microscopic residual disease that is eligible for radical radiotherapy is allowed
  * Patients with completely resected disease who are judged to be at high risk of relapse and who are eligible for radical radiotherapy are allowed

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin ≥ 10 g/dL
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* Must have normal sleeping habits (i.e., normal circadian rhythm)
* Must have had dental assessment and necessary prophylactic dental extractions carried out
* No connective tissue diseases (e.g., systemic lupus, scleroderma, mixed connective tissue disease, rheumatoid arthritis)
* No organic brain syndrome related to chronic alcohol excess or other cause of sufficient severity that would preclude cooperation with treatment
* No active uncontrolled infection
* No history of psychiatric or neurological disorder that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 6 months since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to the head and neck region

Surgery:

* See Disease Characteristics

Other:

* No other concurrent oral hygiene regimen other than that described in the protocol
* No concurrent radioprotective drugs or therapy

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-08-02 (Actual); Primary Completion 2005-03-11 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georg A. Bjarnason, MD, FRCPC, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (14):
- Canada (14):
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Centre at Surrey Memorial Hospital, Surrey, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Regional Cancer Care at Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - McGill Cancer Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bjarnason GA, Mackenzie RG, Nabid A, Hodson ID, El-Sayed S, Grimard L, Brundage M, Wright J, Hay J, Ganguly P, Leong C, Wilson J, Jordan RC, Walker M, Tu D, Parulekar W; National Cancer Institute of Canada Clinical Trials Group (HN3). Comparison of toxicity associated with early morning versus late afternoon radiotherapy in patients with head-and-neck cancer: a prospective randomized trial of the National Cancer Institute of Canada Clinical Trials Group (HN3). Int J Radiat Oncol Biol Phys. 2009 Jan 1;73(1):166-72. doi: 10.1016/j.ijrobp.2008.07.009. Epub 2008 Sep 19. PMID 18805649
- [Result] Bjarnason GA, MacKenzie R, Hodson I, et al.: A randomized prospective phase-III study comparing the acute oral mucositis of morning vs. afternoon radiotherapy (RT) in patients (pts) with squamous cell carcinoma of the head and neck (SCCHN): NCIC-CTG HN.3. [Abstract] J Clin Oncol 23 (Suppl 16): A-LBA5500, 500s, 2005 .